CLINICAL TRIAL: NCT07044609
Title: A Phase IV, Randomized, Placebo-Controlled, Double-Blind Study to Assess the Effectiveness and Safety of Clonidine Extended-Release (OnydaTM XR) in Children Aged 6 to 12 Years With Attention-Deficit/ Hyperactivity Disorder and Oppositional Defiant Disorder
Brief Title: A Study to Assess the Effectiveness and Safety of Clonidine Extended-Release OnydaTM XR in Children With ADHD and ODD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Las Vegas Medical Research, LLC DBA Vector Clinical Trials (Other)
Collaborators: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADHD-01
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Attention-deficit/Hyperactivity Disorder; Oppositional Defiant Disorder in Children
Keywords: ADHD, ODD, oppositional defiant disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, parallel-group study. Subjects will be assigned 1:1 to drug or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clonidine extended-release suspension and placebo suspension look alike. An unblinded pharmacist will dispense the drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Extended-release clonidine oral suspension (Active Comparator): Participants in this arm will start on 0.1 mg of clonidine extended-release oral suspension and titrate to 0.2 mg of clonidine extended release oral suspension.
  Interventions: Drug: Clonidine extended release oral suspension
- Placebo suspension (Placebo Comparator): Participants in this arm will receive a placebo oral-suspension throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine extended release oral suspension — The study is blinded and the active clonidine extended-release oral suspension will look just like the placebo comparator.
  Arms: Extended-release clonidine oral suspension
Drug: Placebo — Placebo suspension
  Arms: Placebo suspension

SUMMARY:
This is a study to see how safe and effective OnydaTM XR is to treat Attention-Deficit/Hyperactivity Disorder (ADHD) in children aged 6 to 12 years who also have Oppositional Defiant Disorder (ODD). The trial will consist of a screening period of up to 28 days; a 35-day double-blind treatment period that includes a one week of the lowest dose of medication (0.1mg) given at bedtime, then three weeks at 0.2 mg, then one week at 0.1 mg and a follow-up phone call one week after stopping study medication. During the screening period, we will determine whether participants qualify to enroll in the study.

Approximately 162 boys and girls aged 6 to 12 years, who are currently diagnosed with ADHD and ODD, are planned to be screened in order to complete approximately 124 subjects.

Key Inclusion/Exclusion Criteria Participants will have a main diagnosis of ADHD and comorbid ODD based on a structured interview. They will also be required to have significant problems because of their ADHD and be in good health. They will not be able to take other medications for ADHD or any other mental health problems during the study.

At the screening visit, participants and their parents will be asked about ADHD, ODD and other mental health symptoms. They will also give blood and urine samples, and complete an electrocardiogram and physical exam. Blood pressure and pulse rate will also be obtained. Parents will complete questionnaires about ADHD, ODD, and sleep.

During the second visit, the doctor will ensure that participants continue to qualify for the study. Parents and participants will complete questionnaires. Parents will be shown how to dose the study medication. It is a liquid suspension.

Participants will be seen weekly and will be asked about changes in health, new medications and parents will complete questionnaires while participants have blood pressure and pulse rate checked.

At the last in-clinic study visit, participants will also have blood and urine samples taken and, complete an electrocardiogram and undergo a physical exam. Parents will complete questionnaires.

One week after the last in-clinic visit

DETAILED DESCRIPTION:
This is a study to see how safe and effective OnydaTM XR is to treat Attention-Deficit/Hyperactivity Disorder (ADHD) in children aged 6 to 12 years who also have Oppositional Defiant Disorder (ODD).

The primary objective of this study is to establish that an optimal dose of OnydaTM XR will result in a significant reduction in attention-deficit/hyperactivity disorder (ADHD) symptoms compared to placebo in children aged 6 to 12 years.

The primary efficacy measure is the change in the ADHD-RS-5 (Investigator Scored) Total Score from Visit 2 (Baseline) to Visit 6 (End of Double-blind Treatment [0.2 mg treatment])

The key secondary objectives include:

* Change on the Conners 4TM Oppositional Defiant Disorder Symptom Scale from Visit 2 to Visit 6
* Change from Visit 2 Baseline to Visit 6 in ADHD-RS-5 Hyperactivity/Impulsivity and Inattention subscale scores

Other secondary measures include:

* Clinical Global Impression Severity Scale change from Visit 2 (Baseline) to Visit 6 (End of Double-blind Treatment [ 0.2 mg treatment])
* Clinical Global Impression Change Scale change from Visit 2 (Baseline) to Visit 6 (End of Double-blind Treatment [ 0.2 mg treatment])
* Children's Sleep Habits Questionnaire (CSHQ)

Safety and tolerability of OnydaTM XR:

* Changes in Blood Pressure, Pulse, Height, and Weight
* Columbia Suicide Severity Rating Scale (C-SSRS)

The trial will consist of a screening period of up to 28 days; a 35-day double-blind treatment period that includes a one week of the lowest dose of medication (0.1mg) given at bedtime, then three weeks at 0.2 mg, then one week at 0.1 mg and a follow-up phone call one week after stopping study medication. During the screening period, we will determine whether participants qualify to enroll in the study.

Approximately 162 boys and girls aged 6 to 12 years, who are currently diagnosed with ADHD and ODD, are planned to be screened in order to complete approximately 124 subjects.

Key Inclusion/Exclusion Criteria Participants will have a main diagnosis of ADHD and comorbid ODD based on a structured interview. They will also be required to have significant problems because of their ADHD and be in good health. They will not be able to take other medications for ADHD or any other mental health problems during the study.

At the screening visit, participants and their parents will be asked about ADHD, ODD and other mental health symptoms. They will also give blood and urine samples, and complete an electrocardiogram and physical exam. Blood pressure and pulse rate will also be obtained. Parents will complete questionnaires about ADHD, ODD, and sleep.

During the second visit, the doctor will ensure that participants continue to qualify for the study. Parents and participants will complete questionnaires. Parents will be shown how to dose the study medication. It is a liquid suspension.

Participants will be seen weekly and will be asked about changes in health, new medications and parents will complete questionnaires while participants have blood pressure and pulse rate checked.

At the last in-clinic study visit, participants will also have blood and urine samples taken and, complete an electrocardiogram and undergo a physical exam. Parents will complete questionnaires.

One week after the last in-clinic visit there will be a phone call to the participant to determine if any adverse events resolved.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 6 to 12 years of age inclusive at time of consent
2. Meets DSM-5 criteria for ADHD, combined, hyperactive/impulsive or inattentive presentation using a clinical interview by an experienced clinician and confirmed with the Mini-International Neuropsychiatric Interview for children and adolescents (MINI-KID)
3. Meets DSM-5 criteria for Oppositional Defiant Disorder confirmed with the MINI-KID
4. The subject has a parent or legal guardian who will give written informed consent for the subject to participate in the study
5. Subject and parent/legal guardian must be able to speak, read, write, and understand English
6. Subject and parent/legal guardian must agree to comply with all protocol requirements
7. ADHD-RS-5 score of ≥28 at Screening and Baseline if not taking ADHD medications. If taking ADHD medication, must have ADHD-RS-5 score of ≥28 after washout at Baseline
8. Subject has a CGI-S score of ≥4 at Screening if not taking ADHD medication. If taking ADHD medication must have CGI-S score of ≥4 at Baseline
9. Subject must live with primary caretaker/rater
10. Sitting systolic and diastolic blood pressure below the 95th percentile for age, gender, and height
11. Subject is functioning at age-appropriate level intellectually based on investigator's opinion
12. If a female has experienced menarche, she must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test at Screening, a negative urine pregnancy test at Baseline, and agree to be abstinent from sexual activity that could result in pregnancy, or use acceptable contraceptives throughout the entire study
13. Must be able to discontinue stimulants 7 days prior to Baseline and nonstimulants 14 days prior to Baseline

Exclusion Criteria:

1. Subject has a current severe comorbid psychiatric condition (except oppositional defiant disorder [ODD]) that is controlled (requiring a prohibited medication or behavioral modification program) or uncontrolled. These conditions include comorbid disorders, such as bipolar illness, psychosis, autism spectrum disorder, post-traumatic stress disorder, obsessive-compulsive disorder, substance use disorder, or conduct disorder, that in the opinion of the Investigator, contraindicate treatment with OnydaTM XR, or confound efficacy or safety assessments
2. Use of another investigational drug in the 30 days prior to screening
3. Use of anticonvulsants, antidepressants, or antipsychotics in the 30 days prior to screening
4. History (in the past 12 months) or presence of clinically significant cardiovascular, cerebrovascular, renal, hepatic, gastrointestinal, pulmonary, immunological, hematological, endocrine, or neurological disease, that in the opinion of the investigator, could put the subject at risk if he/she participates in the trial, or confound study results
5. History of presence of suicidal ideation or self-injurious behavior
6. Subject has orthostatic hypotension or history of hypertension
7. Subject has clinically significant ECG findings as judged by the investigator.
8. Subject has a QTc-Fridericia (QTc-F) > 450 ms in males or > 470 ms in females at screening
9. Subject has participated in another clinical trial within 30 days prior to screening
10. Subject has an allergy or intolerance to clonidine or OnydaTM XR
11. Subject has clinically significant abnormal laboratory values at screening
12. Subject has a positive drug screen at Screening, except for ADHD medications with a valid prescription
13. Subject has a positive drug screen at Baseline
14. Subject is currently considered a suicide risk, has previously made a suicide attempt, or has active suicidal ideation based on the Columbia Suicide Severity Rating Scale. Specifically, any positive response on C-SSRS items 4 or 5 currently at screening, or in the past 12 months, is exclusionary
15. Subject has a history of a seizure disorder, except for children who have had febrile seizures prior to age 5 years
16. Subjects who have been treated with clonidine or guanfacine in the past 30 days
17. History of failure to respond to clonidine or guanfacine
18. Subject started psychotherapy less than 30 days prior to screening

    -

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in the ADHD-RS-5 (Investigator Scored) Total Score from Visit 2 (Baseline) to Visit 6 (End of Double-blind Treatment [0.2 mg treatment]). | 4 weeks
  Change in the ADHD-RS-5 (Investigator Scored) Total Score from Visit 2 (Baseline) to Visit 6 (End of Double-blind Treatment [0.2 mg treatment]).

CONTACTS AND LOCATIONS:
Overall Officials: Ann Childress, MD, Principal Investigator — Vector Clinical Trials

IPD SHARING:
Plan to Share IPD: No
This is a single site study.